CLINICAL TRIAL: NCT00635726
Title: Sequential High Dose MVAC (Methotrexate, Vinblastine, Doxorubicin and Cisplatin), Followed by Gemcitabine Plus Cisplatin in Treating Patients With Locally Advanced or Metastatic Bladder Cancer
Brief Title: Methotrexate, Vinblastine, Doxorubicin and Cisplatin (MVAC) Followed by Gemcitabine Plus Cisplatin (GEM+CDDP) in Locally Advanced or Metastatic Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.16
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Methotrexate; Vinblastine; Doxorubicin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MVAC -> GEM+CDDP
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate intravenous (IV) 30 mgr/m2 on day 1 every 2 weeks for 6 courses
Drug: Vinblastine — Vinblastine IV 3 mgr/m2 on day 1 every 2 weeks for 6 courses
Drug: Doxorubicin — Doxorubicin IV 30 mgr/m2 on day 2 every 2 weeks for 6 courses
Drug: Cisplatin — Cisplatin IV 70 mgr/m2 on day 2 every 2 weeks for 6 courses
  Other Names: CDDP
Drug: Cisplatin — Cisplatin IV 70 mgr/m2 on day 1 every 3 weeks for 4 courses
  Other Names: CDDP
Drug: Gemcitabine — Gemcitabine 1000 mgr/m2 on days 1 and 8 every 3 weeks for 4 courses
  Other Names: Gemzar

SUMMARY:
This phase II trial will study the effectiveness and toxicity of sequential high dose MVAC followed by gemcitabine and cisplatin, as first line treatment in patients with locally advanced or metastatic bladder cancer.

DETAILED DESCRIPTION:
High dose MVAC and Cisplatin/Gemcitabine combination regimens have shown comparable efficacy in the first line treatment of advanced or metastatic bladder cancer, whereas the latter regimen has better tolerability. The efficacy and tolerability of the sequential administration of these two regimens is not known.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell carcinoma of the urinary bladder.
* Metastatic or locally advanced disease.
* No prior chemotherapy.
* Performance status (World Health Organization) 0-2.
* Measurable or evaluable disease.
* Measurable disease is defined as at least 1 unidimensional measurable lesion

  ≥20 mm by conventional techniques or 1 bidimensionally measurable lesion ≥ 20 X 10 mm. Lesions that are smaller or uni- or bidimensionally unmeasurable are considered as evaluable disease.
* Adequate liver (bilirubin ≤ 1.5 Upper Normal Limit, serum glutamate-pyruvate aminotransferase/serum glutamic pyruvic transaminase ≤ 2 Upper Normal Limit, ALP ≤ 2.5 Upper Normal Limit), renal (creatinine ≤ 1.5 Upper Normal Limit) and bone marrow (absolute neutrophil count ≥ 1,500/mm3, platelet count ≥ 100,000/mm3) function.
* Life expectancy > 3 months.
* Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

* History of serious cardiac disease (unstable angina, severe congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias).
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer.
* Active infection.
* Uncontrolled inflammation.
* Pregnant or lactating women.
* Psychiatric illness or social situation that would preclude study compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Objective responses confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Time to tumor progression | 1-year
Overall survival | 1-year
Toxicity profile | Toxicity assessment on each chemotherapy cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Androulakis, MD, Principal Investigator — University Hospital of Crete, Dept. of Medical Oncology
Locations (7):
- Greece (7):
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dept. of Medical Oncology, Athens
  - IASO General Hospital of Athens, 1st Dept. of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Dept. of Internal Medicine, Athens
  - Metaxa's Anticancer Hospital of Piraeus, 1st Dept. of Medical Oncology, Piraeus
  - Theagenion Anticancer Hospital of Thessaloniki, Thessaloniki